CLINICAL TRIAL: NCT07091513
Title: Comparison of Erector Spinae Plane Block, Extrapedicular Infiltration Anesthesia, and Conventional Local Infiltration Anesthesia for Percutaneous Kyphoplasty
Brief Title: Anesthesia for Percutaneous Kyphoplasty
Acronym: Kyphoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Mehmet Burak Eşkin, Associate Professor, Gulhane School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/156
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Vertebral Compression Fracture; Kyphoplasty
Keywords: Kyphoplasty; Vertebral compression fracture; Erector spinae plane block; Local anesthesia

STUDY DESIGN:
Intervention Model Description: A total of 90 ASA I-III patients were randomly assigned into three groups: group CLIA (n=30), group EPIA (n=30), and group ESP (n=30). The same amount of local anesthetic mixture (6 ml lidocaine 1% and 14 ml bupivacaine 0.5%) was used for regional anesthetic techniques in all groups. Fentanyl 0.1 mcg/kg and midazolam 0.1 mg/kg were intravenously (IV) given before prone positioning. Pain was evaluated using Visual Analogue Score (VAS) and sedation level using Ramsay Sedation Scale (RSS) during the procedure. Primary outcome measure were VAS and RSS scores. Secondary outcome measures were hemodynamic changes and additional analgesic and sedative consumptions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group CLIA (Active Comparator): In the CLIA group, the anesthetic needle was angled 10 to 15 degrees with the sagittal plane and was directed towards the laminar periosteum at the pedular projection point in the lamina and a mixture of 1% Lidocaine hydrochloride (6 mL) and 0.5% bupivacaine (14 mL) was injected.
  Interventions: Procedure: group ESP
- Group EPİA (Active Comparator): In the EPIA group, the anesthetic needle was directed towards the lateral half of the pedicle along the lateral superior articular process and the upper border of the transverse process (angulation 5 to 10 degrees with the sagittal plane and 5 to 10 degrees with the coronal plane), followed by the injection of the same 20 mL mixture
  Interventions: Procedure: group ESP
- group ESP (Active Comparator): . In the ESP group, a high frequency linear transducer (HFL50XP, SonoSite Inc., Bothell, WA, USA ) was located vertically approximately 3 cm lateral to the projection point with identification of the spinous process, lamina, transverse process, and the erector spinae muscle. The skin and subcutaneous tissues were infiltrated using 5 mL of 1% Lidocaine Hydrochloride. A 22-G peripheral nerve block needle (50 mm) (SonoTAP, Pajunk, Geisingen, Germany) was inserted in-plane from caudal to cranial between the fascia of the erector spinae muscle and the transverse process under the ultrasound guidance. After hydro-localization using 1 ml of with normal saline, this plane was opened. The same 20 mL mixture of LA was injected after negative aspiration of blood.
  Interventions: Procedure: group ESP

INTERVENTIONS:
Procedure: group ESP — . In the ESP group, a high frequency linear transducer (HFL50XP, SonoSite Inc., Bothell, WA, USA ) was located vertically approximately 3 cm lateral to the projection point with identification of the spinous process, lamina, transverse process, and the erector spinae muscle. The skin and subcutaneous tissues were infiltrated using 5 mL of 1% Lidocaine Hydrochloride. A 22-G peripheral nerve block needle (50 mm) (SonoTAP, Pajunk, Geisingen, Germany) was inserted in-plane from caudal to cranial between the fascia of the erector spinae muscle and the transverse process under the ultrasound guidance. After hydro-localization using 1 ml of with normal saline, this plane was opened. The same 20 mL mixture of LA was injected after negative aspiration of blood.

SUMMARY:
The aim of this study was to compare ESP with conventional local infiltration anesthesia (CLIA) and extrapedicular infiltration anesthesia (EPIA) with respect to analgesic efficacy in patients underwent elective PKP for VCF. A total of 90 ASA I-III patients were randomly assigned into three groups: group CLIA (n=30), group EPIA (n=30), and group ESP (n=30). The same amount of local anesthetic mixture (6 ml lidocaine 1% and 14 ml bupivacaine 0.5%) was used for regional anesthetic techniques in all groups. Fentanyl 0.1 mcg/kg and midazolam 0.1 mg/kg were intravenously (IV) given before prone positioning. Pain was evaluated using Visual Analogue Score (VAS) and sedation level using Ramsay Sedation Scale (RSS) during the procedure. Primary outcome measure were VAS and RSS scores. Secondary outcome measures were hemodynamic changes and additional analgesic and sedative consumptions

DETAILED DESCRIPTION:
Study design This study was conducted as a prospective, single-center, randomized controlled clinical trial in the orthopedic operating rooms of an academic training and research hospital between 26 January 2023 and 31 March 2025 after hospital's ethic committee approval for clinical researches (25.01.2023- protocol no. 2022/156 düzeltme). The trial was registered at ClinicalTrials.gov prior to patient enrollment (NCT04201678). A written informed consent was obtained from all patients participating in the trial. The manuscript adheres to the Consolidated Standards of Reporting Trials (CONSORT) statement. The trial was ended after the pre-planned number of patients who concluded the intended follow-up period. Patients were randomly assigned to one of three parallel groups, initially in 1:1:1 ratio to receive one of the three anesthetic managements for the procedure. The flow diagram is shown in Figure 1.

Participants The American Society of Anesthesiologists (ASA) physical status class I-III patients were included in the study who were between 40 and 85 years and scheduled for an elective, single- level thoracal or lumbar vertebrae kyphoplasty for VCF. The diagnosis was confirmed with physical examination and radiological imaging including direct radiographs, computerized tomography and magnetic resonance imaging. The exclusion criteria were patient refusal, pregnancy, history of previous lumbar surgery, coagulation disorders, anticoagulation medication, abnormal coagulation tests, allergy to the local anesthetics and study drugs, cognitive disorder, chronic pain therapy, and multiple-level vertebrae fractures. It was decided that the patients were dropped out after trial commencement who could not tolerate their position or developed sudden deterioration in vital parameters during the intervention which required emergency treatment. Three staff anesthesiologists and one orthopedic surgeon participated in the study who had more than ten years of experience. Patients were invited on the day before the surgery and a research assistant evaluated the pain of patients at rest using Visual Analogue Scale (VAS) before the procedure.

Patients were randomly assigned to one of three parallel groups in 1:1:1 ratio using the block randomization method. The randomization sequence was developed using a computer-generated table of random groups. Group allocation was concealed using individual sealed opaque envelopes that were numbered in sequential order. As individuals were enrolled in the study, the next envelope in the sequence was extracted and the participant was assigned to the groups accordingly.

All patients were randomly divided into the three study groups that were formed according to anesthesia protocol: 30 patients underwent anesthesia with CLIA, 30 patients with EPIA, and 30 patients with ESP. Patient characteristics including sex, age, weight, height, and basal vital parameters were recorded. Saline or Ringer's lactate solution (1-3 mL.kg-1.h-1, up to 1 L) was intravenously (IV) administered for hydration . In the operating room, the patients were monitored with noninvasive blood pressure (BP), oxygen saturation (SpO2), and electrocardiogram (ECG). Baseline vital parameters were recorded. Patients were given 0.1 mcg/kg fentanyl and 0.1 mg/kg midazolam and carefully positioned to prone on the operation table. Each patient was analyzed with pre-operative and intra-operative VAS scores to evaluate pain perception. Briefly, after explanation of the use of VAS, patients were told that they would be asked to complete the scale at baseline (immediately before surgical preparation) and on the 15th, 20th, 30th and 45th minutes of the surgical procedure. A VAS value of 0 was defined to identify the absence of pain and 10 was defined as maximum pain. Patients with severe pain (defined as a VAS score≥4) received 0.05 mcg/kg fentanyl as an additional analgesic. The sedation levels of patients were evaluated with the Ramsay sedation scale (RSS) at baseline and on the 15th, 20th, 30th and 45th minutes of surgery. The RSS divides a patient's level of sedation into six categories ranging from level 1 (anxious, agitated or restless) to level 6 (deep sedation without any response). The targeted sedation level of patients was RSS 2 or 3. Patients with a sedation score of 1 received additionally 0.05 mg/kg midazolam. Hemodynamic evaluations, including non-invasive measurement of mean arterial BP, heart rate (HR), and SpO2 were monitored at baseline and on the 15th, 20th, 30th and 45th minutes of the surgery. Additional analgesic and sedation amounts applied during the procedures were also recorded.

In CLIA and EPIA groups, the projection point of the pedicle was located as the first step, 5 mL of 1% Lidocaine Hydrochloride was used to infiltrate the skin, subcutaneous tissue and parts of the lumbodorsal muscles, from 1 cm lateral point to pedicle projection point. In the CLIA group, the anesthetic needle was angled 10 to 15 degrees with the sagittal plane and was directed towards the laminar periosteum at the pedular projection point in the lamina and a mixture of 1% Lidocaine hydrochloride (6 mL) and 0.5% bupivacaine (14 mL) was injected. In the EPIA group, the anesthetic needle was directed towards the lateral half of the pedicle along the lateral superior articular process and the upper border of the transverse process (angulation 5 to 10 degrees with the sagittal plane and 5 to 10 degrees with the coronal plane), followed by the injection of the same 20 mL mixture. In the ESP group, a high frequency linear transducer (HFL50XP, SonoSite Inc., Bothell, WA, USA ) was located vertically approximately 3 cm lateral to the projection point with identification of the spinous process, lamina, transverse process, and the erector spinae muscle. The skin and subcutaneous tissues were infiltrated using 5 mL of 1% Lidocaine Hydrochloride. A 22-G peripheral nerve block needle (50 mm) (SonoTAP, Pajunk, Geisingen, Germany) was inserted in-plane from caudal to cranial between the fascia of the erector spinae muscle and the transverse process under the ultrasound guidance. After hydro-localization using 1 ml of with normal saline, this plane was opened. The same 20 mL mixture of LA was injected after negative aspiration of blood.

The primary outcome measure was pain (VAS) scores. The secondary outcome measures were additional rescue analgesics.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status class I-III patients
* 40 -85 years old
* Elective, single- level thoracal or lumbar vertebrae kyphoplasty for VCF

Exclusion Criteria:

* patient refusal
* pregnancy,
* history of previous lumbar surgery,
* coagulation disorders,
* anticoagulation medication
* abnormal coagulation tests,
* allergy to the local anesthetics and study drugs,
* cognitive disorder,
* chronic pain therapy
* multiple-level vertebrae fractures

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-01-26 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
VAS scores | Briefly, after explanation of the use of VAS, patients were told that they would be asked to complete the scale at baseline (immediately before surgical preparation) and on the 15th, 20th, 30th and 45th minutes of the surgical procedure.
  A VAS value of 0 was defined to identify the absence of pain and 10 was defined as maximum pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Gülhane Medical Faculty, Ankara, KEÇiören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided